CLINICAL TRIAL: NCT03426332
Title: Management of Adrenal Emergency in Germany - a Prospective Multicenter
Brief Title: Management of Adrenal Emergency in Germany
Acronym: MAdEy
Status: Completed | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: University Hospital, Frankfurt, Germany (Unknown); Endocrinology in Charlottenburg, Berlin, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: MAdEy-Study
Record Dates: First submitted 2018-01-18; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Adrenal Insufficiency
Keywords: Adrenal Insufficiency; Adrenal crisis; Adrenal emergency; Glucocorticoid injection
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The management of adrenal crisis is often problematic and the time to adequate treatment is frequently delayed.The aim of the study is to evaluate the management of adrenal emergencies requiring parenteral glucocorticoid treatment by a prospective multicenter study in patients with chronic adrenal insufficiency.

DETAILED DESCRIPTION:
Despite established hormone replacement therapy, patients with chronic adrenal insufficiency (AI) are at risk of suffering from adrenal crisis (AC). Further data suggests that the management of AC is often problematic and the time to adequate treatment is frequently delayed.The aim of the study is to evaluate the management of adrenal emergencies (AE) requiring parenteral glucocorticoid (GC) treatment by a prospective multicenter study.

Patients with chronic AI receive a questionnaire on the management of emergency situations, which had to be completed and sent back in case of an emergency requiring parenteral GC administration. Furthermore, patients were contacted by phone in case of a missing response every six months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Documented chronic adrenal insufficiency
* Established corticosteroid replacement therapy
* Written informed consent

Exclusion Criteria:

- Age <18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years with a documented chronic adrenal insufficiency under established corticosteroid replacement therapy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Median time from contacting a medical professional to arrival of professional medical help | 6-36 months
  Evaluation of the median time (in minutes) from contacting a medical professional (by the patient) to arrival of professional medical help during an (adrenal) emergency.
  The time is documented in a questionnaire by the patients themselves (directly after the adrenal emergency). The data of all patients will be stated as median and range.
Median time from showing the emergency card (by a patient) to glucocorticoid-injection by a medical professional | 6-36 months
  Evaluation of the median time (in minutes) from showing the emergency card (by a patient) to glucocorticoid-injection by a medical professional.
  The time is documented in a questionnaire by the patients themselves (directly after the adrenal emergency). The data of all patients will be stated as median and range.
Median time from the beginning of symptoms to glucocorticoid-injection | 6-36 months
  Evaluation of the median time (in minutes) from the beginning of symptoms to glucocorticoid-injection during an (adrenal) emergency.
  The time is documented in a questionnaire by the patients themselves (directly after the adrenal emergency). The data of all patients will be stated as median and range.
Duration of hospitalisation (number of days at a hospital) | 6-36 months
  Evaluation of the duration of hospitalisation (number of days at a hospital) due to an adrenal emergency.
  The number of days is documented by the patients themselves (directly after the adrenal emergency). The data of all patients will be stated as median and range.
Number of patients that received an intramuscular glucocorticoid-injection | 6-36 months
  Evaluation of the number of patients that received an intramuscular glucocorticoid-injection (compared to subcutaneous administration) during an adrenal emergency. Documentation by the patients themselves directly after the adrenal emergency.

SECONDARY OUTCOMES:
Cause of the adrenal emergency | 6-36 months
  Evaluation of the causes of the adrenal emergencies. The causes are documented in a questionnaire by the patients themselves. The number of different causes that are stated by all patients will be evaluated.
Median time from the beginning of symptoms to oral dose adjustment (glucocorticoids) during an adrenal emergency | 6-36 months
  Evaluation of the median time (in minutes) from the beginning of symptoms to oral dose adjustment (glucocorticoids).
  The time is documented in a questionnaire by the patients themselves (directly after the adrenal emergency). The data of all patients will be stated as median and range.
Median time from the beginning of symptoms to contacting a medical professional | 6-36 months
  Evaluation of the median time (in minutes) from the beginning of symptoms to contacting a medical professional during an adrenal emergency.
  The time is documented in a questionnaire by the patients themselves (directly after the adrenal emergency). The data of all patients will be stated as median and range.
Symptoms of the adrenal emergency | 6-36 months
  Evaluation of the symptoms during the adrenal emergencies. The symptoms are documented in a questionnaire by the patients themselves. The number of different symptoms that are stated by all patients will be evaluated.
Median amount of additionally oral ingested glucocorticoids during the adrenal emergency | 6-36 months
  Evaluation of the median amount of additionally oral ingested glucocorticoids (in mg) during the adrenal emergency.
  The amount of glucocorticoids is documented in a questionnaire by the patients themselves (directly after the adrenal emergency). The data of all patients will be stated as median and range.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hahner S, Spinnler C, Fassnacht M, Burger-Stritt S, Lang K, Milovanovic D, Beuschlein F, Willenberg HS, Quinkler M, Allolio B. High incidence of adrenal crisis in educated patients with chronic adrenal insufficiency: a prospective study. J Clin Endocrinol Metab. 2015 Feb;100(2):407-16. doi: 10.1210/jc.2014-3191. Epub 2014 Nov 24. PMID 25419882
- [Background] Hahner S, Hemmelmann N, Quinkler M, Beuschlein F, Spinnler C, Allolio B. Timelines in the management of adrenal crisis - targets, limits and reality. Clin Endocrinol (Oxf). 2015 Apr;82(4):497-502. doi: 10.1111/cen.12609. Epub 2014 Nov 6. PMID 25200922
- [Background] Allolio B. Extensive expertise in endocrinology. Adrenal crisis. Eur J Endocrinol. 2015 Mar;172(3):R115-24. doi: 10.1530/EJE-14-0824. Epub 2014 Oct 6. PMID 25288693